CLINICAL TRIAL: NCT06386666
Title: A Prospective, Multicenter, Single-group, Target-value Clinical Trial to Evaluate the Safety and Efficacy of Single-use Annular Sutures for Annular Incisions Following Nucleus Pulposus Removal
Brief Title: A Clinical Trial to Evaluate the Safety and Efficacy of Single-use Fibrous Ring Sutures for the Suture of Fibrous Ring Incision After Nucleus Pulposus Removal
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Suzhou Kerui Medical Technology Co., Ltd (Other)
Collaborators: 2020 (Beijing) Medical Technology Co., Ltd (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: RLRL-CTP
Record Dates: First submitted 2024-04-15; First posted 2024-04-26 (Actual); Last update posted 2024-07-19 (Actual); Status verified 2024-07

CONDITIONS: Intervertebral Disc Disorder
MeSH Terms: conditions — Intervertebral disc disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- The fibrous ring was sutured using a disposable fibrous ring suturing device (Experimental)
  Interventions: Device: Disposable fibrous ring sutures

INTERVENTIONS:
Device: Disposable fibrous ring sutures — A new disposable fibrous ring suture device developed and produced by 2020 (Beijing) Medical Technology Co., Ltd

SUMMARY:
The objective of this clinical trial was to evaluate the safety and effectiveness of single-use annular sutures for the closure of annular incisions after nucleus pulposus removal. Participants used single-use annular sutures to close the annular fibers. The success rate of suture, reduction value of annulus, proportion of annulus reduction, intraoperative blood loss, suture time, VAS pain score (low back, bilateral lower extremities), Oswestry index (ODI index), and Short were evaluated The effectiveness evaluation results of Form-12 health survey (SF-12 score), treatment success rate, device defects, product operation satisfaction, and safety evaluation results of recurrence rate, adverse events, and serious adverse events were used to verify the safety and effectiveness of disposable fibrillar suture for annular incision suture after nucleus pulposus removal.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years old, gender unlimited;
2. Meet the diagnosis of lumbar disc herniation (refer to the Guidelines for Diagnosis and Treatment of Lumbar disc herniation), and expect to undergo single-level disc nucleus pulposus extraction;
3. The history of lumbar disc herniation is more than 6 weeks, and systematic conservative treatment is ineffective；
4. ODI index ≥20 points;
5. In the VAS score of bilateral lower limbs, at least one side was ≥4 points;
6. The score of the three evaluation indicators according to the modified Pfirrmann grade, age and disc height is no more than 7 points (see Annex 1 for the criteria);
7. Voluntarily participate and sign informed consent;
8. Be able to communicate well with research doctors, have good compliance, and can follow the requirements of clinical research.

Exclusion Criteria:

1. Laboratory examination (blood routine examination, blood biochemistry, coagulation function and blood pregnancy, etc.), imaging examination (MRI) and vital signs examination have abnormal results with clinical significance, and the researchers believe that they are not suitable for inclusion;
2. Active local or systemic infection;
3. Patients with lumbar tumors and/or spinal malformations;
4. Imaging showed calcification of the posterior longitudinal ligament;
5. A history of serious diseases of important organs (such as cardiovascular system, liver, lung, kidney and nervous system);
6. There are autoimmune diseases or abnormal coagulation function;
7. Previous or planned surgical procedures to fuse or stabilize the lumbar spine during the trial;
8. Intraoperative exploration of the location of the annulus fibriatus could not satisfy the requirement that the needle entry point was more than 2mm away from the margin of the annulus fibriatus;
9. Pregnant or lactating women, or those who have a pregnancy plan during the trial period;
10. Those who are participating in other clinical trials at the same time;
11. Other situations that the researcher considers inappropriate to participate in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Estimated)
Dates: Start 2024-08-15 (Estimated); Primary Completion 2025-08-29 (Estimated); Study Completion 2025-11-15 (Estimated)

PRIMARY OUTCOMES:
Success rate of suture | Immediately after surgery
  After the intraoperative suture was completed, the quality of the suture was evaluated by the investigator. After all subjects completed the operation, the success rate of suture was calculated.
  Evaluation criteria: 1) No sutures fell off during the suture process; 2) No suture fracture during the suture process; 3) A sterile scale was used to measure annulus fibrosus cleft before and after suture, and medical image data were retained. Finally, the size changes of cleft before and after suture were compared. The size of the wound after suture should be reduced by more than 60% compared with that before suture (the size of the annulus fibrous tear should be determined by its maximum diameter).
  If all the above three conditions are met, the suture is successful. If any one of the conditions is not met, the suture is failed.
  Successful rate of suture = Number of successful sutures/total number of sutures *100%

SECONDARY OUTCOMES:
Annulus fibril cleft decreased in value | During the surgery.
  The change of annulus cleft was evaluated according to annulus suture.Annular cleft reduction = annular cleft size before suture - annular cleft size after suture.
Reduced proportion of annular fibril cleft | During the surgery.
  The change of annular tear reduction was assessed according to annular suture.Annulus cut reduction ratio = (size of annulus cut before unsutured - size of annulus cut after sutured)/size of annulus cut without suture *100%
Intraoperative blood loss | The day after the surgery
  Information on intraoperative blood loss was obtained from surgical records.
Suture time | The day after the surgery
  The time between assembly and completion of the suture from the single use of the ring suture.
Treatment success rate | Six months after surgery
  After the subjects completed the 6-month post-operation interview, the researchers made the judgment. If the subjects met all the following evaluation criteria, they were recorded as "treatment success"; otherwise, they were "treatment failure".Evaluation criteria: 1) ODI index decreased by ≥10 points compared with pre-operation; 2) Compared with the preoperative results, the VAS score of lower extremities decreased by ≥2 points (if only one side was ≥4 points, that side was dominant; If both sides are ≥4 points, the average score of both sides is used to calculate the VAS score decline value); 3) No nerve root symptoms; 4) No second operation and/or other therapeutic intervention at the treated site after surgery; 5) MRI images showed no swelling or other abnormalities of clinical significance in the operative segment.
  Treatment success rate = Number of successful cases/total cases *100%
VAS pain score (lower back, bilateral lower limbs) | Before surgery, 4 days after surgery, 1 month after surgery, 3 months after surgery, 6 months after surgery
  According to their subjective feelings, the subjects were evaluated by Visual Analogue Scales (VAS). On a 10cm scale, "0" means painless and "10" means the most intense pain.
SF-12 rating | Before surgery, 4 days after surgery, 1 month after surgery, 3 months after surgery, 6 months after surgery
  The SF-12 Health Questionnaire consists of 12 questions divided into 2 dimensions: physical health and mental health. Each question is set with different options, subjects according to their own feelings and actual situation, choose the most suitable option, each option corresponds to a different score. The score ranges from 0 to 100, with higher scores indicating better physical and mental health, and lower scores indicating worse physical and mental health.
ODI index | Before surgery, 4 days after surgery, 1 month after surgery, 3 months after surgery, 6 months after surgery
  ODI index includes 3 areas of single function, pain and individual comprehensive function, with a total of 10 items, the score range is 0 ~ 5 points, the total score is 50 points, the higher the score, the more serious the dysfunction of the subject.

OTHER OUTCOMES:
Recurrence rate | From the day of surgery to 6 months after surgery
  The relapses of the subjects were closely observed and recorded by the researchers. If radiculopathy occurs and the MRI shows that the disc at the original surgical level has herniated again and is pressing on the nerve tissue, it can be considered a "recurrence." Recurrence rate = Number of recurrence cases/total cases ×100%.